CLINICAL TRIAL: NCT01351610
Title: Open, Randomized, Mono-Centre, Two-Parallel Group Clinical Phase I/II Trial on the Evaluation of Tolerability and Efficacy of an Intravenous Infusion of Human Bone Marrow Derived Autologous, CD34-Negative Mesenchymal Stem Cells for the Treatment of Critical Limb Ischemia in Patients With Advanced Peripheral Arterial Occlusive Disease Subsequent to Percutaneous Transluminal Angioplasty
Brief Title: Tolerability and Efficacy of Intravenous Infusion of Autologous MSC_Apceth for the Treatment of Critical Limb Ischemia
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Apceth GmbH & Co. KG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MSC_Apceth_001
Record Dates: First submitted 2011-05-10; First posted 2011-05-11 (Estimated); Last update posted 2015-12-15 (Estimated); Status verified 2015-12

CONDITIONS: Critical Limb Ischemia; Peripheral Artery Disease
Keywords: Critical Limb Ischemia; Peripheral Arterial Occlusive Disease; Peripheral Artery Disease; Peripheral Vascular Disease; Stem Cell Therapy; Mesenchymal Stem Cells
MeSH Terms: conditions — Chronic Limb-Threatening Ischemia; Peripheral Arterial Disease; Peripheral Arterial Occlusive Disease 1; Peripheral Vascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group B (Experimental)
  Interventions: Procedure: PTA
- Group A (Experimental)
  Interventions: Biological: PTA + Infusion of MSC_Apceth

INTERVENTIONS:
Biological: PTA + Infusion of MSC_Apceth — percutaneous transluminal angioplasty followed by infusion of MSC_Apceth
  Arms: Group A
Procedure: PTA — percutaneous transluminal angioplasty only
  Arms: Group B

SUMMARY:
MSC_Apceth are GMP-manufactured, autologous ex-vivo expanded non-hemapoietic bone-marrow derived stem cells for the treatment of Critical Limb Ischemia

ELIGIBILITY:
Inclusion Criteria:

1. Patients with peripheral arterial occlusive disease (symptomatic PAOD), diagnosis of CLI defined as persistent, recurring ischemic rest pain for at least 2 weeks, and/or ulceration or gangrene of the foot or toe, with an ABPI </= 0.5,
2. Patients with staging of ≥III according to Fontaine and ≥4 according to Rutherford categories,
3. Patients fulfilling the criteria for an invasive re-vascularisation procedure (PTA) at the discretion of the investigator,
4. Patients without major amputation of the lower extremities within the period of 6 months after inclusion in the opinion of the investigator,

Exclusion Criteria:

1. Patients with wounds of a severity of greater than grade 2 on the Wagner Scale,
2. Patients with life-threatening ventricular arrhythmia,
3. Patients with unstable angina pectoris,
4. Patients with severe congestive heart failure (i.e. NYHA Stage IV),
5. Patients with uncontrolled hypertension (defined as diastolic blood pressure >110 mmHg or systolic blood pressure >180 mmHg during screening),
6. Patients with an uncontrolled diabetes mellitus (HbA1c > 9%),
7. Patients having any history of malignant tumour in the anamnesis or are currently on tumour treatment,
8. Patients who are unsuitable for a MSC stem cell therapy in the opinion of the investigator,

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2011-03; Primary Completion 2014-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Collection of adverse events | one year
Safety laboratory values | 1 year
ECG findings | 1 year
Analysis of inflammation markers | 1 year

SECONDARY OUTCOMES:
Comparison of course of haemodynamic and vascular processes | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Peter Heider, MD, PhD, Principal Investigator — Isar Medizin Zentrum, München
Locations (1):
- Isar Medizin Zentrum, Munich, Bavaria, Germany